CLINICAL TRIAL: NCT00718653
Title: Effects of Antioxidants on Human Macular Pigments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Kyung-Jin Yeum, Tufts Univeristy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: R03EY015674 (NIH); R03EY015674 (NIH)
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-02

CONDITIONS: Eye Health
Keywords: Macular pigment, lutein, green tea extract, antioxidant
MeSH Terms: interventions — Lutein; Tea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): lutein
  Interventions: Dietary Supplement: Lutein
- 2 (Experimental): Lutein plus green tea extract
  Interventions: Dietary Supplement: Lutein plus green tea extract

INTERVENTIONS:
Dietary Supplement: Lutein — Lutein (12 mg/d)
  Arms: 1
Dietary Supplement: Lutein plus green tea extract — lutein (12 mg/d) plus green tea extract (200 mg/d)
  Arms: 2

SUMMARY:
Age-related macular degeneration (AMD) is the leading cause of blindness in the United States. Low dietary intake or low blood levels of lutein and zeaxanthin, which are the only pigments found in the macular region of the human retina, has been associated with an increased risk for AMD. We have reported that the dietary supplementation of lutein and zeaxanthin can increase the macular pigments (MP) of the eye. MP effectively absorbs blue light as well as quenches reactive oxygen species (ROS). Green tea polyphenols are also effective scavenger of ROS in vitro.

Our goal is to elucidate how to effectively increase MP by physiologic levels of antioxidant supplementation. We hypothesize that lutein and tea polyphenols protect the macula of the eye by increasing MP carotenoids effectively through an antioxidant mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Normal hematologic parameters, normal serum albumin, normal liver function, normal kidney function, absence of fat malabsorption and no drug intake which would interfere with fat absorption, metabolism or blood clotting
* non-smokers

Exclusion Criteria:

* A history of kidney stones, active small bowel disease or resection, atrophic gastritis, hyperlipidemia, insulin-requiring diabetes, alcoholism, pancreatic disease, or bleeding disorders
* Exogenous hormone users
* weighing greater than 20% above or below the NHANES median standard
* subjects with serum lutein/zeaxanthin concentrations that are more than 150 % of median of normal population (as previously reported in NHANES III at same age group)
* early age related macular degeneration, cataract, or glaucoma except for those with age appropriate progression of the eye status.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
macular pigments, Plasma lutein concentrations | Every month - baseline, 1, 2, 3, & 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Jin Yeum, Ph.D., Principal Investigator — Tufts Medical Center
Locations (1):
- Jean Mayer USDA-Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Result] Li L, Duker JS, Yoshida Y, Niki E, Rasmussen H, Russell RM, Yeum KJ. Oxidative stress and antioxidant status in older adults with early cataract. Eye (Lond). 2009 Jun;23(6):1464-8. doi: 10.1038/eye.2008.281. Epub 2008 Sep 19. PMID 18806766
- See also: Related Info — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?cmd=Retrieve&db=PubMed&dopt=Citation&list_uids=18806766